CLINICAL TRIAL: NCT06579690
Title: Effectiveness and Safety Dosing of Sodium Bicarbonate in Women With Obstructed Labor in Eastern Uganda: A Phase III Randomized Placebo-controlled Trial
Brief Title: Use of Preoperative Sodium Bicarbonate Among Women With Obstructed Labor
Acronym: SoBicOL-II
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Busitema University (Other)
Collaborators: University of Liverpool (Other); Oslo University Hospital (Other); Cures Within Reach (Other); Open Philanthropy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BusitemaU2
Record Dates: First submitted 2024-08-27; First posted 2024-08-30 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Obstructed Labor
Keywords: Sodium bicarbonate; Obstructed labor; Women; Uganda
MeSH Terms: conditions — Dystocia | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 8.4g of 8.4% sodium bicarbonate solution Arm (Experimental): Each participant will receive 100mls of 8.4g, 8.4% sodium bicarbonate solution, up to two doses, four hours apart.
  Interventions: Drug: 8.4% sodium bicarbonate solution
- 12.6g of 8.4% sodium bicarbonate solution Arm (Experimental): Each participant will receive 150mls of 12.6g, 8.4% sodium bicarbonate solution, up to two doses, four hours apart.
  Interventions: Drug: 8.4% sodium bicarbonate solution
- 16.8g of 8.4% sodium bicarbonate solution Arm (Experimental): Each participant will receive 200mls of 16.8g, 8.4% sodium bicarbonate solution, up to two doses, four hours apart.
  Interventions: Drug: 8.4% sodium bicarbonate solution
- Normal Saline 0.9% Arm (Active Comparator): Each participant will receive 50mls of Normal Saline 0.9%, up to two doses, four hours apart.
  Interventions: Other: 0.9% Normal Saline

INTERVENTIONS:
Drug: 8.4% sodium bicarbonate solution — Sodium bicarbonate infusion 8.4% solution The study drug will be contained in identical 25 mL glass vials (Neon Laboratories Ltd, Mumbai, India), administered intravenously as a single bolus dose.
  Arms: 12.6g of 8.4% sodium bicarbonate solution Arm; 16.8g of 8.4% sodium bicarbonate solution Arm; 8.4g of 8.4% sodium bicarbonate solution Arm
Other: 0.9% Normal Saline — The comparision group will receive 50 mls of 0.9% Normal Saline
  Arms: Normal Saline 0.9% Arm

SUMMARY:
The goal of this clinical trial is to determine a universal safe and effective dose of sodium bicarbonate for use among women with Obstructed labour to treat acidosis. It will also learn about the safety of sodium bicarbonate drug among women with Obstructed labour.

Researchers will compare sodium bicarbonate drug to normal saline (a look-alike solution) to see if sodium bicarbonate works to treat acidosis.

Participants will receive sodium bicarbonate solution or a placebo up to two doses, four hours apart.

DETAILED DESCRIPTION:
Oral bicarbonate is a safe, cheap and effective acid buffer, widely used in sports to improve performance because of its ability to prevent and reverse the effects of metabolic acidosis. Clinically, it is used in intensive care units to treat patients with overwhelming infections or poisoning. In low resource settings, obstructed labor (OL) is a major problem that accounts for 22% of maternal deaths. The fetal harm of OL comes from intrapartum asphyxia, characterized by accumulation of hydrogen ions that cross the placental barrier to cause fetal acidosis. Acidosis causes failure of basic cellular functions resulting into cell death. In a recent Randomised Clinical Trial, the investigators found that 61% of 477 women with OL were acidotic (lactate >4.8 mmol/L), with a median capillary blood lactate level of 6.9 (3.4-13) mmol/L.

The investigators propose an early phase III, placebo-controlled dose-ranging trial to determine the efficacy and safety of a pre-operative infusion of sodium bicarbonate in women with obstructed labour (OL). In a ratio of 1:1:1: 1 100 mls (8.4g), 150 mls (12.6g) and 200 mls (16.8g) of 8.4% sodium bicarbonate solution, or placebo (50 mls of Normal Saline 0.9%). The primary outcome will be mean change in acidosis (pH and lactate levels) from baseline. The secondary outcomes will be neonatal death, safety of sodium bicarbonate, pharmacokinetics of sodium bicarbonate in pregnant women, primary postpartum haemorrhage, sepsis, and maternal death.

ELIGIBILITY:
Inclusion Criteria:

* Patients with obstructed labour
* Must be a singleton pregnancy
* Must be a term pregnancy (≥37 weeks of gestation)
* Must be in cephalic presentation.

Exclusion Criteria:

* Patients with other obstetric emergencies such as antepartum haemorrhage, preeclampsia and eclampsia (defined as elevated blood pressure of at least 140/90 mm Hg, urine protein of at least 2+, any of the danger signs and fits), premature rupture of membranes and intrauterine fetal death.
* Patients with comorbidities such as diabetes mellitus, sickle cell disease, renal disease, liver disease and heart disease.
* Patients with hypokalaemia (148 mmol/L) and alkalosis (bicarbonate >22 mmol/L) because they are more likely to develop adverse drug reactions

Ages: 16 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 280 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Mean change in maternal pH from baseline in each group | At baseline, 30, 60, 90, 120 and 150 minutes
Mean umbilical blood pH in each arm of the study | At baseline, 30, 60, 90, 120 and 150 minutes

SECONDARY OUTCOMES:
Mean lactate in maternal and umbilical blood, | At baseline and at birth.
Number of early neonatal deaths | Within 7 days
Safety of sodium bicarbonate (comparison of the proportion of participants that get side effects in each arm) | Within 24 hours after administration of the drug
Number of mothers that get primary postpartum hemorrhage | Within 24 after birth

CONTACTS AND LOCATIONS:
Overall Officials: Trond Michelsen, PhD, Principal Investigator — Oslo University Hospital; David Mukunya, PhD, Principal Investigator — Busitema University; Julius Wandabwa, PhD, Principal Investigator — Busitema University; Kenneth Mugabe, MD, Principal Investigator — Busitema University; Dan Kibuule, PhD, Principal Investigator — Busitema University; Andrew Weeks, MD, Principal Investigator — University of Liverpool

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be freely available.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Immediately following publication, No end date
Access Criteria: Anyone who wishes to access the data. Any types of data analyses will be permitted.